CLINICAL TRIAL: NCT04975321
Title: A Clinical Trial of NuSmile's Pre-Veneered Stainless Steel Crowns and NuSmile ZR Crowns Compared With Strip Composite Crowns in Anterior Primary Teeth -- Pilot Study
Brief Title: Clinical Trial NuSmile Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Mariella Garcia, Associate Professor, School of Dentistry: Dept. of Pediatric Dentistry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003980
Record Dates: First submitted 2021-06-01; First posted 2021-07-23 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: Primary Dental Caries, Multisurface Origin (Diagnosis)
Keywords: Anterior primary teeth restorations
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Nu Smile Zirconia crown (Active Comparator): Anterior primary teeth which received a NuSmile zirconia crown as a final restoration
  Interventions: Device: Nu Smile Zirconia crown
- Nu Smile pre veneered crown (Active Comparator): Anterior primary teeth which received a NuSmile pre veneered crown as a final restoration
  Interventions: Device: Nu Smile Pre Veneered crown
- Composite strip crown (Active Comparator): Anterior primary teeth which received a composite strip crown as a final restoration
  Interventions: Device: Composite strip crown

INTERVENTIONS:
Device: Nu Smile Zirconia crown — Placement of an anterior primary crown restoration
  Arms: Nu Smile Zirconia crown
Device: Nu Smile Pre Veneered crown — Placement of an anterior primary crown restoration
  Arms: Nu Smile pre veneered crown
Device: Composite strip crown — Placement of an anterior primary crown restoration
  Arms: Composite strip crown

SUMMARY:
A clinical trial comparing two types of NuSmile anterior crowns to composite strip crowns on anterior dental restorations.

DETAILED DESCRIPTION:
Stainless steel crowns have been the most common treatment for large cavities in baby teeth until recently. These crowns are silver in color, and aesthetically are not a good option for restoring front teeth. Several tooth colored options have been developed to meet the growing demand for more aesthetics on front teeth. With the variety of new options for restoring anterior primary teeth, the investigators would like to evaluate the long-term success of three tooth-colored restoration options: NuSmile Signature crowns, NuSmile ZR crowns, and composite crowns. The investigators are interested in looking at the outcomes of these three restoration types, in terms of durability, aesthetics and cost effectiveness for the treatment of front baby teeth. The purpose of this pilot study is to evaluate the clinical performance of two types of NuSmile crowns compared to composite crowns in treating large multi-surfaced cavities on front baby teeth.

ELIGIBILITY:
Inclusion Criteria:

* Patients of record at the University of Washington's Center for Pediatric Dentistry
* Patients in general good health (ASA I)
* Patients aged 5 years old or younger
* Patients in need of at least one preformed crowns, on anterior primary teeth
* Patients undergoing general anesthesia for dental treatment
* Parent or guardian of patient able and willing to provide informed consent

Exclusion Criteria:

* Medically compromising condition
* Teeth with proximal space closures of sufficient magnitude to preclude placement of crown
* Teeth with complete absence of facial or lingual walls following tooth preparation
* Teeth that are expected to be exfoliated/extracted within one year will not participate in the study
* Anterior crowding
* Occlusion class III

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 97 (Actual)
Dates: Start 2015-06-06 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2019-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariella Garcia, DDS, Principal Investigator — University of Washington
Locations (1):
- University of Washington-The Center for Pediatric Dentistry, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment start date was 06/05/2015 and last day was 10/16/2018 . All recruitment took place at the The Center for Pediatric Dentistry
Pre-assignment Details: Initial enrollment was performed at the time of dental consent before general anesthesia procedure for all patients. Once the patient enrolled and consented to participate they will be evaluated clinically for remaining inclusion and exclusion criteria during the general anesthesia procedure. 21 patients were not meeting inclusion criteria or met the exclusion criteria so form 97 patients that were enrolled only 76 patients were allocated in the different arms of the study
Units Other Than Participants: teeth
Period: Overall Study
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Started | 25; 70 teeth | 26; 80 teeth | 25; 70 teeth
Completed | 15; 40 teeth | 15; 47 teeth | 17; 48 teeth
Not Completed | 10; 30 teeth | 11; 33 teeth | 8; 22 teeth

BASELINE CHARACTERISTICS:
Units Other Than Participants: teeth
Groups:
- Total: Total of all reporting groups
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown | Total
Number analyzed (Participants) | 15 | 15 | 17 | 47
Number analyzed (teeth) | 40 | 47 | 48 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 17 | 47
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.4 (0.8) | 3.4 (0.8) | 3.4 (0.8) | 3.4 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 9 | 26
  Male | 9 | 4 | 8 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0
    (all) |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 17 | 76

OUTCOME MEASURES:

1. Primary Outcome: Fitting
Description: The number of teeth scored in the crown fitting categories described below
  Fitting 0 = Good natural retention
  1. Moderate natural retention
  2. Little or no natural retention
  A higher score means a worse outcome
Time Frame: 12 months
Population: Number of teeth analyzed per group
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Number analyzed (Participants) | 15 | 15 | 17
Number analyzed (Teeth) | 40 | 47 | 48
Teeth
  0= Good retention | 37 | 42 | 48
  1=Moderate natural retention | 3 | 5 | 0

2. Primary Outcome: Positioning
Description: Change in the following clinical assessment measure between baseline and 12 months using the categories below
  Positioning
  0= Proper position
  1. Rotated - in occlusion
  2. Not in occlusion with or without rotation
  A higher score means a worse outcome
Time Frame: 12 months
Population: Number of teeth analyzed per group
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Number analyzed (Participants) | 15 | 15 | 17
Number analyzed (Teeth) | 40 | 47 | 48
Teeth
  Proper position | 40 | 45 | 46
  Rotated- in occlusion | 0 | 2 | 2

3. Primary Outcome: Proximal Contact
Description: The number of teeth scored in the proximal contact categories as described below
  Proximal contact 0= Open spaces
  1. Floss meets little or no resistance when passes through contact
  2. Floss meets significant when passes through contact
  A higher score means a worse outcome
Time Frame: 12 months
Population: Number of teeth analyzed per group
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Number analyzed (Participants) | 15 | 15 | 17
Number analyzed (Teeth) | 40 | 47 | 48
Teeth
  Open spaces | 30 | 41 | 44
  Floss meets little or no resistance when passes through contact | 9 | 6 | 4
  Floss meets significant when passes through contact | 1 | 0 | 0

4. Primary Outcome: Marginal Adaptation
Description: The number of teeth scored in the marginal adaptation categories as described below
  Marginal adaptation 0= No discrepancies detected with explorer
  1. Detectable discrepancies but clinically acceptable
  2. Detectable discrepancies, not acceptable -replacement required
  A higher score means a worse outcome
Time Frame: 12 months
Population: Number of teeth analyzed per group
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Number analyzed (Participants) | 15 | 15 | 17
Number analyzed (Teeth) | 40 | 47 | 48
Teeth
  No discrepancies detected with explorer | 40 | 47 | 43
  Detectable discrepancies but clinically acceptable | 0 | 0 | 5

5. Primary Outcome: Color
Description: The number of teeth scored in the color categories described below
  Color matching
  0= Matches completely or within range of shade and translucency
  1. Outside range for yellow, yellow/brown discoloration or gray discoloration
  2. Outside range for reason other than yellowing or graying
  A higher score means a worse outcome
Time Frame: 12 months
Population: Number of teeth analyzed per group
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Number analyzed (Participants) | 15 | 15 | 17
Number analyzed (Teeth) | 40 | 47 | 48
Teeth
  Matches completely or within range of shade and translucency | 40 | 47 | 48
  Outside range for yellow, yellow/brown discoloration or gray discoloration | 0 | 0 | 0

6. Primary Outcome: Gingival Status
Description: The number of teeth scored in the gingival status categories described below
  Gingival status 0=Pink, firm, free of inflammation
  1. Red and/or inflamed - no bleeding on probing
  2. Spontaneous and excessive bleeding on probing
  A higher score means a worse outcome
Time Frame: 12 months
Population: Number of teeth analyzed per group
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Number analyzed (Participants) | 15 | 15 | 17
Number analyzed (Teeth) | 40 | 47 | 48
Teeth
  Pink, firm, free of inflammation | 9 | 5 | 0
  Red and/or inflamed - no bleeding on probing | 8 | 18 | 14
  Spontaneous and excessive bleeding on probing | 23 | 24 | 34

7. Primary Outcome: Retention of the Crown
Description: The number of teeth scored in the retention of the crown categories described below
  Retention of the crown 0= Intact
  1= Partially missing 2 = Missing - some cement remaining on both tooth and crown interior
  A higher score means a worse outcome
Time Frame: 12 months
Population: Number of teeth analyzed per group
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Number analyzed (Participants) | 15 | 15 | 17
Number analyzed (Teeth) | 40 | 47 | 48
Teeth
  Intact | 40 | 47 | 48
  Partially missing | 0 | 0 | 0

8. Primary Outcome: Integrity of the Veneer/Composite
Description: The number of teeth scored in the integrity of the veneer/composite categories described below
  Integrity of veneer/ composite 0= Intact
  1. Partially missing - one third missing
  2. Completely missing
  A higher score means a worse outcome
Time Frame: 12 months
Population: Number of teeth analyzed per group
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Number analyzed (Participants) | 15 | 15 | 17
Number analyzed (Teeth) | 40 | 47 | 48
Teeth
  Intact | 40 | 47 | 47
  Partially missing - one third missing | 0 | 0 | 1

9. Primary Outcome: Secondary Caries
Description: The number of teeth scored in the secondary caries categories described below
  Secondary caries 0= Absent
  1= Present
  A higher score means a worse outcome
Time Frame: 12 months
Population: Number of teeth analyzed per group
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Number analyzed (Participants) | 15 | 15 | 17
Number analyzed (Teeth) | 40 | 47 | 48
Teeth
  Absent | 39 | 43 | 42
  Present | 1 | 4 | 6

10. Primary Outcome: History of Trauma
Description: The number of teeth scored in the history of trauma categories described below
  History of trauma 0= Absent
  1= Present
  A higher score means a worse outcome
Time Frame: 12 months
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Number analyzed (Participants) | 15 | 15 | 17
Number analyzed (Teeth) | 40 | 47 | 48
Teeth
  Absent | 39 | 38 | 47
  Present | 1 | 9 | 1

11. Primary Outcome: Clinical Pulp Pathology
Description: The number of teeth scored in the clinical pulp pathology categories described below
  Clinical pulp pathology 0= Absent
  1= Present
  A higher score means a worse outcome
Time Frame: 12 months
Population: Number of teeth analyzed per group
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Number analyzed (Participants) | 15 | 15 | 17
Number analyzed (Teeth) | 40 | 47 | 48
Teeth
  Absent | 39 | 47 | 47
  Present | 1 | 0 | 1

12. Primary Outcome: Radiographical Pulp Pathology
Description: The number of teeth scored in the radiographical pulp pathology categories described below Radiographical pulp pathology 0= Absent
  1= Present A higher score means a worse outcome A higher score means a worse outcome
Time Frame: 12 months
Population: Number of teeth analyzed per group
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Number analyzed (Participants) | 15 | 15 | 17
Number analyzed (Teeth) | 40 | 47 | 48
Teeth
  Absent | 37 | 43 | 48
  Present | 3 | 4 | 0

13. Primary Outcome: Parent's Esthetic Satisfaction
Description: The number of teeth scored in the parent's esthetic satisfaction categories described below
  Parents esthetic satisfaction via a survey 0=Satisfied
  1= Dissatisfied
  A higher score means a worse outcome
Time Frame: 12 months
Population: Number of teeth analyzed per group
Measure: Count of Units; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
Number analyzed (Participants) | 15 | 15 | 17
Number analyzed (Teeth) | 40 | 47 | 48
Teeth
  Satisfied | 38 | 47 | 48
  Dissatisfied | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: No reports of adverse events in all three groups
Arm/Group | Nu Smile Zirconia Crown | Nu Smile Pre Veneered Crown | Composite Strip Crown
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/17

LIMITATIONS AND CAVEATS:
Many families had moved, changed or lost phone services, or were otherwise unable to be reached. There were also a few families who withdrew following treatment due to a disinterest in travelling the distance for follow-up care. The loss of follow up was similar for all treatment groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-11-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT04975321/Prot_SAP_000.pdf
  • Informed Consent Form (2015-06-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT04975321/ICF_001.pdf